CLINICAL TRIAL: NCT05049460
Title: Adjunctive Transcranial Stimulation to Reduce Impulsivity in Opiate Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56570
Record Dates: First submitted 2021-09-08; First posted 2021-09-20 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Opioid-use Disorder; Tobacco Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active intervention (Active Comparator): Four sessions of theta burst stimulation, amounting to 7200 pulses at 120% resting motor threshold. Targeting will be done using neuronavigation and processed resting state brain scan.
  Interventions: Device: Theta Burst Stimulation
- Sham TMS (Placebo Comparator): Four sessions of sham TMS. Targeting will be done using neuronavigation and processed resting state brain scan.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Theta Burst Stimulation — Four sessions of theta burst stimulation (TBS) at 120 % RMT and comprising 7200 pulses, given with functional targeting.
  Arms: Active intervention
Device: Sham TMS — Four sessions of sham TMS, done using the A/P MagVenture coil, with subject's head separated from the coil by foam padding.
  Arms: Sham TMS

SUMMARY:
The goal of this study is to examine the effect of four sessions of theta burst stimulation (TBS) versus sham TMS on attentional bias for smoking and opioid cues versus neutral stimuli in a population of patients with tobacco use disorder (TUD) with comorbid opioid use disorder (OUD) that is stable and on treatment with buprenorphine. The investigators will also examine the effect of TBS on craving for cigarettes as well as opioids. Participants will perform a stress induction procedure that mirrors an optimum combination of cues that trigger tonic craving in their environment while exposed to stress. All four sessions of TBS/sham TMS will be performed on the same day, with each session lasting for approximately 10 minutes and separated by 50 minute intervals.

DETAILED DESCRIPTION:
Tobacco use disorder (TUD) is highly comorbid with opioid use disorder (OUD). Craving in TUD as well as OUD is of two kinds - phasic and tonic. Phasic craving is present at baseline and tonic craving is accentuated by environmental stimuli. A predominant mediator of tonic craving is attentional bias (AB) for environmental stimuli related to either smoking or opioid use.

The study is comprised of two days of participation. On the first day, participants will perform two attentional bias (AB) paradigms - one to assess their baseline AB for smoking cues versus neutral cues and another AB paradigm to assess baseline AB for opioid cues versus neutral cues. Craving will be assessed using tobacco craving questionnaire and a visual analogue scale (for opioids), in the context of participants performing a stress induction procedure (which will be a combination of the cold pressor test and PASAT). The investigators will also acquire a baseline resting state fMRI in addition to MRPAGE structural T1 and T2W sequences.

On the second day, participants will receive either four sessions of TBS or sham TMS. Targeting will be down using processed resting state brain scan. Each session of TBS or sham TMS will last approximately 10 minutes. During each of the 50 minute intervals between stimulation sessions, participants will perform AB paradigms for smoking and opioids. The craving scale with stress induction will be performed twice - once before the sessions and once after the four sessions of TBS/sham TMS. The investigators will also acquire resting state scans after the four sessions of TBS/sham TMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the SMART Clinic at University of Kentucky
* 18-60 years of age
* Preferably right hand dominant
* Currently self-report smoking 10 of more cigarettes per day or a score of > 5 on the Fagerstrom Test for Nicotine
* Willing and able to abstain from all drug use
* Exhaled breath on day of study CO < 10 ppm
* Stabilized on maintenance buprenorphine if having comorbid opioid use disorder
* Able to read and speak English
* Able to provide informed consent to participate.

Exclusion Criteria:

* Pregnant, nursing, or becoming pregnant during the study.
* History of traumatic brain injury or seizures which are contraindications for transcranial magnetic stimulation (TMS).
* Increased risk of seizure for any reason, including prior diagnosis of epilepsy, seizure disorder, increased intracranial pressure, or history of significant head trauma with loss of consciousness for ≥ 5 minutes which are all contraindications for TMS.
* Presence of intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes), cardiac pacemakers, or vagus nerve stimulation device which are all contraindications for magnetic resonance imaging.
* Neurological disorder including, but not limited to: space occupying brain lesion; any history of seizures, history of cerebrovascular accident; fainting, cerebral aneurysm, major neurocognitive disorder, Huntington chorea; multiple sclerosis which are all contraindications for TMS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rush, PhD, Study Chair — Professor, Department of Behavioral Sciences
Locations (1):
- 245 Fountain Court, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rakesh G, Alcorn JL 3rd, Khanal R, Himelhoch SS, Rush CR. Comparing cigarette-cue attentional bias between people with HIV/AIDS and people with opioid use disorder who smoke. Health Psychol Behav Med. 2023 Sep 7;11(1):2255028. doi: 10.1080/21642850.2023.2255028. eCollection 2023. PMID 37693107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Intervention | Sham TMS
Started | 12 | 11
Completed | 8 | 7
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Sham TMS | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.13 (10.97) | 35.43 (5.16) | 36.87 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Attentional Bias for Smoking Stimuli
Description: Attentional bias was measured at baseline using a visual probe task administered (adapted for smoking images) on a computer and an eye tracker. Images of cigarettes and matched neutral images were presented on a laptop screen, 3 cm apart. Upon offsetting the image pairs, a visual probe (X) appeared on either the left or right side of the screen, in the exact location of one of the previously presented images. Attentional bias is quantified by subtracting the average fixation time on neutral cues from the average fixation time on cigarette cues. The fixation time is measured with an eye tracker in milliseconds.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
milliseconds | 501.53 (145.24) | 406.70 (116.41)

2. Primary Outcome: Attentional Bias for Smoking Stimuli
Description: Attentional bias was measured using a visual probe task administered (adapted for smoking images) on a computer and an eye tracker. Images of cigarettes and matched neutral images were presented on a laptop screen, 3 cm apart. Upon offsetting the image pairs, a visual probe (X) appeared on either the left or right side of the screen, in the exact location of one of the previously presented images. Attentional bias is quantified by subtracting the average fixation time on neutral cues from the average fixation time on cigarette cues. The fixation time is measured with an eye tracker in milliseconds.
Time Frame: Immediately after intervention (sessions of TBS or sham TMS)
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
milliseconds | 275.83 (158.14) | 414.52 (254.3)

3. Primary Outcome: Attentional Bias for Opioid Stimuli
Description: Attentional bias was measured using a visual probe task administered (adapted for opioid images) on a computer and an eye tracker. Images of opioids and matched neutral images were presented on a laptop screen, 3 cm apart. Upon offsetting the image pairs, a visual probe (X) appeared on either the left or right side of the screen, in the exact location of one of the previously presented images. Attentional bias is quantified by subtracting the average fixation time on neutral cues from the average fixation time on opioid cues. The fixation time is measured with an eye tracker in milliseconds.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
milliseconds | 373.09 (176.06) | 132.01 (70.89)

4. Primary Outcome: Attentional Bias for Opioid Stimuli
Description: as for outcome 3
Time Frame: Immediately after intervention (sessions of TBS or sham TMS)
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
milliseconds | 305.80 (196.95) | 158.61 (198.75)

5. Primary Outcome: Craving
Description: The Tobacco Craving Questionnaire-short form (TCQ-SF) consists of 12 items rated on a visual analogue scale from 0 to 84 with a higher score equating to increased craving.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
units on a scale | 57.8 (5.3) | 53.1 (6.1)

6. Primary Outcome: Craving
Description: as for outcome 5
Time Frame: Immediately after intervention (sessions of TBS or sham TMS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 8 | 7
units on a scale | 54.1 (6.3) | 48.7 (4.9)

7. Secondary Outcome: Number of Participants Showing Functional Connectivity Changes
Description: Changes in resting state network changes caused by TBS/sham TMS
Time Frame: Baseline and immediately after intervention (sessions of TBS or sham TMS)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Intervention | Sham TMS
Number analyzed (Participants) | 7 | 7
Participants | 7 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events were reported
Arm/Group | Active Intervention | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT05049460/Prot_ICF_001.pdf